CLINICAL TRIAL: NCT03298815
Title: A Randomized, Double-Blinded, Placebo-Controlled Study for the Treatment of Ocular Chronic Graft-Versus-Host Disease (GVHD) With Amniotic Fluid Eye Drops (AFED)
Brief Title: Study for the Treatment of Ocular Chronic Graft-Versus-Host Disease (GVHD) With Amniotic Fluid Eye Drops (AFED)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Catherine Lee, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103515
Record Dates: First submitted 2017-09-13; First posted 2017-10-02 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Ocular Graft Versus Host Disease
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amniotic Fluid Eye Drops (AFED) - All participants, One eye (Active Comparator)
  Interventions: Biological: Amniotic Fluid Eye Drops (AFED)
- Saline Solution - All participants, One eye (Placebo Comparator)
  Interventions: Other: Saline Solution

INTERVENTIONS:
Biological: Amniotic Fluid Eye Drops (AFED) — One drop (0.25 mL) in one eye twice daily for up to 3 months
  Arms: Amniotic Fluid Eye Drops (AFED) - All participants, One eye
Other: Saline Solution — One drop (0.25 mL) in the other eye twice daily for up to 3 months
  Arms: Saline Solution - All participants, One eye

SUMMARY:
A Randomized, Double-blinded, Placebo-Controlled Study for the Treatment of Ocular Chronic Graft Verses Host Disease with Processed Amniotic Fluid (pAF) Drops.

DETAILED DESCRIPTION:
This is a randomized (to each eye, within patient), double-blinded, placebo-controlled study of the efficacy of Processed Amniotic Fluid (pAF) in patients with hematologic malignancies who have undergone Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) and are diagnosed with Chronic Graft Verses Host Disease of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed within 5 years after hematopoietic stem cell transplant for any disease, with any graft and any conditioning regimen with at least one of the following symptoms:

  1. Dry eye symptoms partially affecting (requiring lubricant drops > 3 x per day or punctal plugs, or thermally cauterized puncta) or significantly affecting (special eyeware to relieve pain) activities of daily living (ADL)
  2. Unable to work because of ocular symptoms
  3. Loss of vision due to keratoconjunctivitis sicca (KCS)
* Patients may be using bilateral scleral lenses and/or bilateral punctal plugs at the time of accrual.
* Patients who are 18 years of age or older.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Patients who have any other reversible cause for dry eye at the time of accrual.
* More than 3 lines of therapy beyond corticosteroids with or without calcineurin inhibitors or sirolimus
* Relapsed malignancy at time of accrual after the most recent transplantation
* A difference in dryness between both eyes of more than 2 points of the grading provided by the International Dry Eye Workshop (DEWS) 2007 report
* Patients who are pregnant or plan to become pregnant while participating in the study.
* Patients who are not willing to discontinue the use of any eye drops, with the exception of non-medicated lubricant eye drops (artificial tears). All eye drops (excluding non-medicated lubricant eye drops) must be stopped at least seven days before treatment with pAF.
* Inability to comply with the investigational plan and visit schedule for any reason, in the judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Lee, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Amniotic Fluid Eye Drops (AFED): Subjects received both Amniotic Fluid Eye Drops and Saline Solution. One eye was randomized to receive amniotic fluid drops and the other eye received saline solution drops.
  Amniotic Fluid Eye Drops (AFED): One drop (0.25 mL) in one eye twice daily for up to 3 months
- Saline Solution: Subjects received both Amniotic Fluid Eye Drops and Saline Solution. One eye was randomized to receive amniotic fluid drops and the other eye received saline solution drops.
  Saline Solution: One drop (0.25 mL) in the other eye twice daily for up to 3 months
Period: Overall Study
Arm/Group | Amniotic Fluid Eye Drops (AFED) | Saline Solution
Started | 15; 15 eyes | 15; 15 eyes
Completed | 15; 15 eyes | 15; 15 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects received both Amniotic Fluid Eye Drops and Saline Solution. Each were randomized to one eye.
  Amniotic Fluid Eye Drops (AFED): One drop (0.25 mL) in one eye twice daily for up to 3 months Saline Solution: One drop (0.25 mL) in the other eye twice daily for up to 3 months
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Baseline Functional Assessment of Cancer Therapy - General (FACT-G) Score [Median (Full Range); unit: units on a scale] — The FACT-G is a 27-item patient-reported questionnaire used to assess the impact of cancer therapy on quality of life. The questionnaire has 5-point Likert scale ranging from 0 (not at all) to 4 (very much) for every question. Questions are added together for an overall score. Higher scores represent better quality of life (range from 0 to 108).
  units on a scale | 88 [58 to 103.8]
Subject wears contacts (scleral lenses) [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response is a composite of the NIH Consensus Conference (CC) for assessment of response in chronic GVHD (eye score) and the International Dry Eye Workshop (DEWS) grading scale. Responders would be defined as a one point improvement in the dry eye grading scale (DEWS), without worsening in the eye score.
Time Frame: 30 days
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Amniotic Fluid Eye Drops (AFED) - All Participants, One Eye | Saline Solution - All Participants, One Eye
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
eyes | 3 | 6
Statistical Analysis 1: Comparison: Amniotic Fluid Eye Drops (AFED) - All Participants, One Eye vs Saline Solution - All Participants, One Eye; Test type: Superiority; p = 0.375, McNemar

2. Secondary Outcome: Change in Functional Assessment of Cancer Therapy: General (FACT-G) From Baseline to 30 Days
Description: Change in Quality of Life questionnaire from baseline to 30 days. FACT-G is a combination score of physical, social/family, emotional, and functional well-being. The score ranges from 0 to 108. The higher the score, the better the quality of life.
Time Frame: baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: Change in score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 15
Change in score on a scale | -1 [-6 to 2.7]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.391, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Functional Assessment of Cancer Therapy: General (FACT-G) From Baseline to 60 Days
Description: Change in Quality of Life questionnaire from baseline to 60 days. FACT-G is a combination score of physical, social/family, emotional, and functional well-being. The score ranges from 0 to 108. The higher the score, the better the quality of life.
Time Frame: baseline and 60 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 15
score on a scale | 2.8 [-1.8 to 3.2]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.267, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy: General (FACT-G) From Baseline to 100 Days
Description: Change in Quality of Life questionnaire from baseline to 100 days. FACT-G is a combination score of physical, social/family, emotional, and functional well-being. The score ranges from 0 to 108. The higher the score, the better the quality of life.
Time Frame: baseline and 100 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 15
score on a scale | 3.0 [-4.0 to 10.3]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.445, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in National Institutes of Health (NIH) Consensus Criteria (CC) Ocular Score of Chronic GVHD From Baseline to 30 Days
Description: Change in ocular score using a four-point scale from 0 (no dry eye symptoms) to 3 (severe dry eye symptoms) from baseline to 30 days.
Time Frame: baseline and 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 13
Participants
  Better results for pAF eye vs Placebo eye | 3
  Better results for Placebo eye vs pAF eye | 0
  Same Directional Results for Both Eyes | 10
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.250, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in National Institutes of Health (NIH) Consensus Criteria (CC) Ocular Score of Chronic GVHD From Baseline to 60 Days
Description: Change in ocular score using a four-point scale from 0 (no dry eye symptoms) to 3 (severe dry eye symptoms).
Time Frame: baseline and 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
Participants
  Better results for pAF eye vs. Placebo eye | 1
  Better results for Placebo eye vs pAF eye | 0
  Same Directional Results for Both Eyes | 14
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 1.00, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in National Institutes of Health (NIH) Consensus Criteria (CC) Ocular Score of Chronic GVHD From Baseline to 100 Days
Description: Change in ocular score using a four-point scale from 0 (no dry eye symptoms) to 3 (severe dry eye symptoms).
Time Frame: baseline and 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
Participants
  Better results for pAF eye vs Placeob eye | 2
  Better results for Placebo eye vs pAF eye | 0
  Same Directional Results for Both Eyes | 13
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.500, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Dry Eye Workshop (DEWS) 2007 Dry Eye Severity Grading From Baseline to 30 Days
Description: Ophthalmologic assessment to determine changes in dry eye signs/symptoms each graded on a scale of 1 to 4 with 1 being non/mild to 4 being most severe for a total score.
Time Frame: baseline and 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 13
Participants
  Better results for pAF eye vs Placebo eye | 3
  Better results for Placebo eye vs pAF eye | 5
  Same Directional Results for Both Eyes | 5
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.563, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Dry Eye Workshop (DEWS) 2007 Dry Eye Severity Grading From Baseline and 60 Days
Description: as for outcome 8
Time Frame: baseline and 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  Better results for pAF eye vs Placebo eye | 0
  Better results for Placebo eye vs pAF eye | 8
  Same Directional Results for Both eyes | 6
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Dry Eye Workshop (DEWS) 2007 Dry Eye Severity Grading From Baseline and 100 Days
Description: as for outcome 8
Time Frame: baseline and 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 13
Participants
  Better results for pAF eye vs Placebo eye | 1
  Better results for Placebo eye vs pAF eye | 5
  Same Directional Results for Both Eyes | 7
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.156, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Pain Assessment From Baseline to 60 Days
Description: Change in patient reported pain level per treatment eye using 0-10 pain rating scale with zero being no pain to 10 being very severe pain. Each individual pain score was used to estimate a regression slope for each eye with pain as the outcome and day of pAF treatments as the explanatory variable.
Time Frame: baseline and 60 days
Measure: Median (Inter-Quartile Range); unit: regression slope
Arm/Group | Amniotic Fluid Eye Drops (AFED) - All Participants, One Eye | Saline Solution - All Participants, One Eye
Number analyzed (Participants) | 15 | 15
regression slope | -0.004 [-0.029 to 0.019] | -0.010 [-0.021 to 0.009]
Statistical Analysis 1: Comparison: Amniotic Fluid Eye Drops (AFED) - All Participants, One Eye vs Saline Solution - All Participants, One Eye; Test type: Superiority; p = 0.208, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Changes in Visual Acuity
Description: Ophthalmologic assessment to determine changes in visual acuity related to the administration of pAF.
Time Frame: baseline, 30 days, 60 days, and 100 days
Population: One participant at the 30 day and 100 day visit did not complete visual acuity assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  Change from baseline to 30 days: number analyzed (Participants) | 13
  Change from baseline to 30 days: Better results for pAF eye vs Placebo eye | 5
  Change from baseline to 30 days: Better results for Placebo eye vs pAF eye | 2
  Change from baseline to 30 days: Same directional results for both eyes | 6
  Change from baseline to 60 days: Better results for pAF eye vs Placebo eye | 2
  Change from baseline to 60 days: Better results for Placebo eye vs pAF eye | 5
  Change from baseline to 60 days: Same directional results for both eyes | 7
  Change from baseline to 100 days: number analyzed (Participants) | 13
  Change from baseline to 100 days: Better results for pAF eye vs Placebo eye | 3
  Change from baseline to 100 days: Better results for Placebo eye vs pAF eye | 2
  Change from baseline to 100 days: Same directional results for both eyes | 8
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.594, Wilcoxon (Mann-Whitney) — 30 day visit
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority; p = 0.469, Wilcoxon (Mann-Whitney) — 60 day visit
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority; p = 0.750, Wilcoxon (Mann-Whitney) — 100 day visit

13. Secondary Outcome: Effects on the Corneal Surface
Description: Ophthalmologic assessment to determine the effects of treatment with pAF on the corneal surface of patients with ocular chronic GVHD.
Time Frame: Up to 100 days
Population: A participant missed the 30 day visit and another missed the 100 day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  30 day visit: number analyzed (Participants) | 13
  30 day visit: Better results for pAF eye vs Placebo eye | 1
  30 day visit: Better results for Placebo eye vs pAF eye | 7
  30 day visit: Same directional results for both eyes | 5
  60 day visit: Better results for pAF eye vs Placebo eye | 3
  60 day visit: Better results for Placebo eye vs pAF eye | 4
  60 day visit: Same directional results for both eyes | 7
  100 day visit: number analyzed (Participants) | 13
  100 day visit: Better results for pAF eye vs Placebo eye | 0
  100 day visit: Better results for Placebo eye vs pAF eye | 3
  100 day visit: Same directional results for both eyes | 10
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.063, Wilcoxon (Mann-Whitney) — 30 day visit
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority; p < 1.000, Wilcoxon (Mann-Whitney) — 60 day visit
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority; p = 0.250, Wilcoxon (Mann-Whitney) — 100 day visit

ADVERSE EVENTS:
Time Frame: Adverse Events are collected through the whole duration of the trial through day 100.
Arm/Group | Amniotic Fluid Eye Drops (AFED) - All Participants, One Eye | Saline Solution - All Participants, One Eye
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amniotic Fluid Eye Drops (AFED) - All Participants, One Eye (N=15) | Saline Solution - All Participants, One Eye (N=15)
Eye Disorders (Eye disorders) | 1 (1) | 1 (1)
Eye disorders (Eye disorders) | 1 (1) | 0 (0) — Eye inflammation
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0) — Application site pain

LIMITATIONS AND CAVEATS:
Main limitation of this study was the randomization of eyes within subjects as some had mild asymmetric disease between eyes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03298815/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT03298815/SAP_002.pdf
  • Informed Consent Form (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT03298815/ICF_003.pdf